CLINICAL TRIAL: NCT03223155
Title: A Randomized Phase I Trial to Evaluate Concurrent Or Sequential Ipilimumab, Nivolumab, and Stereotactic Body Radiotherapy in Patients With Stage IV Non-Small Cell Lung Cancer (COSINR Study)
Brief Title: Concurrent or Sequential Immunotherapy and Radiation Therapy in Patients With Metastatic Lung Cancer
Acronym: COSINR
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-0547
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Stage IV Small Cell Lung Cancer
Keywords: Small cell lung cancer; ipilimumab; nivolumab; stereotactic body radiotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Nivolumab; Ipilimumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequential Arm (Experimental): Patients will be randomized to either the Sequential Arm or the Concurrent Arm. Patients in the Sequential Arm will complete SBRT to 2-4 sites and then begin treatment with nivolumab/ipilimumab between 1-7 days after completion of SBRT.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Radiation: Stereotactic body radiation therapy
- Concurrent Arm (Experimental): Patients will be randomized to either the Sequential Arm or the Concurrent Arm. Patients in the Concurrent Arm will begin treatment with nivolumab/ipilimumab first and must complete planned SBRT to 2-4 sites within 2 weeks (prior to second dose of nivolumab).
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Radiation: Stereotactic body radiation therapy

INTERVENTIONS:
Drug: Nivolumab — Patients in Sequential Arm will begin treatment with nivolumab (given with ipilimumab) between 1-7 days after completion of SBRT.
  Patients in Concurrent arm will begin treatment with nivolumab (given with ipilimumab) first and will continue treatment within 2 weeks, after completion of SBRT to 2-4 sites.
  In both arms, patients will receive treatment with nivolumab 3 mg/kg as a 30-minute infusion +/- 10 minutes every 2 weeks for a maximum of 24 months. Patients will receive treatment on days 1, 15, and 29 of each 6 week cycle.
  Other Names: Opdivo
Drug: Ipilimumab — Patients in Sequential Arm will begin treatment with ipilimumab (given with nivolumab) between 1-7 days after completion of SBRT.
  Patients in Concurrent arm will begin treatment with ipilimumab (given with nivolumab) first and will continue treatment within 2 weeks, after completion of SBRT to 2-4 sites.
  In both arms, patients will receive treatment with ipilimumab 1 mg/kg as a 30-minute +/- 10 minutes infusion every 6 weeks for a maximum of 24 months. Patients will receive treatment on day 1 of each 6 week cycle.
  Other Names: Yervoy
Radiation: Stereotactic body radiation therapy — All patients will receive 3 or 5 fractions of radiation as determined by the location of the lesions to be irradiated. There should be a minimum of 40 hours between treatments for an individual lesion. However, a patient may receive radiation for different lesions on consecutive days. Starting dose depends on metastasis locations.
  Other Names: SBRT

SUMMARY:
Trial Design

* Patients with stage IV non-small cell lung cancer are randomized to nivolumab/ipilimumab plus either sequential or concurrent stereotactic body radiotherapy (SBRT).
* The primary endpoint is the phase I safety endpoint of SBRT dose for each body site.
* The same starting SBRT dose levels are used in each arm. If two or more patients experience a dose-limiting toxicity (DLT) at the starting dose level, then the reduced dose level will be used (Section 7.1-Page 72).
* DLT is defined as any grade ≥3 toxicity possibly, likely, or definitely related to SBRT plus nivolumab/ipilimumab (the combination and not the individual components).
* Irradiated metastases will be grouped into one of five locations, which have different SBRT doses, and the DLTs will be attributed to the relevant organ system.
* The starting and decreased SBRT dose levels are found in Table 2 (Page 20).
* SBRT will be delivered in 3-5 fractions over the course of 1-1.5 weeks.
* Patients in the sequential arm will begin immunotherapy between 1-7 days after completion of SBRT
* Given the accrual data for IRB15-1130, the investigators anticipate that approximately 1/3 of patients will contribute metastasis to 2 locations. Since there are 2 arms, and 5 metastasis locations with 6 patients per location for the starting dose level, this translates to 40 patients for the starting dose level, and another 40 patients should each of the 5 locations require de-escalation to the lower dose level.
* Secondary endpoints include comparisons of efficacy and toxicity between the arms, as well as interrogation of changes in the immune microenvironment induced by the two approaches.

ELIGIBILITY:
Inclusion Criteria:

* 1. Have a histologic diagnosis of stage IV NSCLC.
* 2. Be willing and able to provide written informed consent/assent for the trial.
* 3. Be greater than or equal to 18 years of age on day of signing informed consent.
* 4. Have measurable disease based on RECIST 1.1 including at least two metastatic lesions that meet criteria for SBRT radiation.

  a. 0.25 cc to 65 cc of viable tumor (i.e. primary disease or metastases) approximately 5cm in maximal dimension. Tumors larger than 65 cc can be partially treated
* 5. For biopsy identified patients: Be willing to undergo repeat biopsy of a target lesion before treatment and after radiation. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may be exempted from this requirement after consultation with the Principal Investigator.
* 6. Have a performance status of 0 or 1 on the ECOG Performance Scale.
* 7. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.

Table 1 Adequate Organ Function Laboratory Values System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥ 1,500 /mcL Platelets ≥ 100,000 / mcL Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)

Renal Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤ 1.5 X upper limit of normal (ULN) OR ≥ 50 mL/min for subject with creatinine levels > 1.5 X institutional ULN

Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases Albumin ≥ 3.0 mg/dL aCreatinine clearance should be calculated per institutional standard.

* 8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 24hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* 9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* 10. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* 11. Have an investigator determined life expectancy of at least 6 months.
* 12. Patients whose tumors known to harbor an exon 19 deletion or exon 21 L858R EGFR mutation must have progressed on or had intolerance to an EGFR TKI. Patients whose tumors are known to harbor an ALK translocation must have progressed on or had intolerance to an ALK inhibitor.

Exclusion Criteria:

* 1. Has received prior chemotherapy for NSCLC with the exception of neoadjuvant or adjuvant platinum-based chemotherapy for NSCLC completed >6 months prior to enrollment.
* 2. Has prior exposure to anti-PD1/PD-L1 or anti-CTLA4 therapy.
* 3. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* 4. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy at a dose of >10mg prednisone daily or equivalent at time of first dose of trial treatment.
* 5. Has a known history of active TB (Bacillus Tuberculosis).
* 6. Hypersensitivity to nivolumab, ipilimumab, or any of its excipients.
* 7. Has received radiation therapy within 2 weeks of study drug administration.
* 8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* 9. Patients with untreated symptomatic brain metastases. Patients with treated brain metastases will be allowed if brain imaging obtained greater than 7 days from treatment reveals stable disease. Patients with small (< 3mm) asymptomatic brain metastasis are allowed to enroll. Patients on steroids doses higher than 10 mg of prednisone (or its equivalent) are excluded.
* 10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* 11. Has known history of non-infectious pneumonitis that required steroids or active pneumonitis.
* 12. Has evidence of interstitial lung disease.
* 13. Has an active infection requiring systemic therapy.
* 14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* 15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* 16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* 17. If known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected) then patient is not eligible for cohorts including SBRT to liver lesions.
* 18. Has received a live vaccine within 30 days of planned start of study therapy.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

* 19. Has had prior radiation therapy (defined as >10% of prior prescription dose) to the area planning to be treated with SBRT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of serious adverse events | Up to 4 years
  To determine the recommended SBRT dose to various metastatic locations in patients with stage IV NSCLC when delivered prior to or concurrently with nivolumab and ipilimumab.

SECONDARY OUTCOMES:
Number of adverse events of grade 3-4 or higher | Up to 4 years
  To estimate and compare rates of ≥ grade 3-4 adverse events, by organ system, by CTCAEv4.0 that occur within 3 months from the start of SBRT when given prior to or concurrently with nivolumab/ipilimumab.
Rate of long term adverse events | Up to 4 years
  To estimate and compare the rates of long-term adverse events (after 3 months) from the end of SBRT when given prior to or concurrently with nivolumab/ ipilimumab.
Rate of response | From the start of treatment until the date of first documented progression or date of death from any cause, whichever comes first, up to 100 months
  Summarize and compare the response rate to determine the progression-free survival at 6 months with SBRT given either prior to or concurrently with nivolumab/ipilimumab.
Rate of lesion control | Up to 4 years
  To determine and compare the control of lesion(s) (SBRT treated and non-treated) when given either prior to or concurrently with nivolumab/ipilimumab.
Rate of change in tumor microenvironment | Up to 4 years
  To evaluate and compare changes in the tumor microenvironment induced by radiation when given prior to or concurrently with nivolumab/ipilimumab.
Rate of PD-L1 expression levels response | Up to 4 years
  To evaluate whether response to therapy correlates with PD-L1 expression levels among patients treated with nivolumab/ipilimumab either concurrently or sequential to SBRT.
Measure of peripheral blood cell T cell levels | From the start of treatment, not to exceed 4 years
  To explore whole PBMC by measuring peripheral blood cell T cell subset IFNγ ELISPOT levels throughout the study course and correlate with response to treatment.
Quantification of T cell receptor | From the start of treatment until the date of first documented progression or date of death from any cause, whichever comes first, up to 100 months
  To explore peripheral blood T cell receptor deep sequencing quantification of T cell receptor (TCR) repertoire changes throughout the study course and how TCR repertoire may correlate with progression free survival and/or overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Chmura, MD, PhD, Study Chair — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States